CLINICAL TRIAL: NCT06809920
Title: Analysis of Knee Joint Stability, Functional Capacity, Postural Control, Activation and Muscle Strength of Patients with Anterior Cruciate Ligament Injury Undergoing Physiotherapy After Two Different Surgical Techniques: a Randomized Clinical Trial.
Brief Title: Analysis of Knee Joint of Patients with Anterior Cruciate Ligament Injury Undergoing Physiotherapy After Two Different Surgical Techniques: a Randomized Clinical Trial.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual de Londrina (Other)
Responsible Party: Principal Investigator, Christiane Macedo, Principal Investigator PhD, Universidade Estadual de Londrina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6.955.081
Record Dates: First submitted 2025-01-11; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Anterior Cruciate Ligament (ACL) Tear; Anterior Cruciate Ligament Reconstruction Rehabilitation
Keywords: Knee; Knee Injuries; Anterior Cruciate Ligament Reconstruction; Physiotherapy
MeSH Terms: conditions — Lacerations; Knee Injuries

STUDY DESIGN:
Intervention Model Description: Participants will undergo, in a previously randomized manner, two surgical techniques for reconstruction of the anterior cruciate ligament of the knee. The two techniques differ in the preparation of the graft. Group 1: ACL reconstruction surgery with the conventional technique or, Group 2: Conventional reconstruction surgery of the Anterior Cruciate Ligament + Reconstruction of the Anterolateral Ligament of the knee. The literature indicates that both techniques have good results, but the differences during the rehabilitation process are still unknown. Both groups will be evaluated and reevaluated in the same way. Also, both groups will undergo the same rehabilitation protocol with manual therapy, physical resources (heat, cold, electrotherapy), kinesiotherapy, and isokinetic exercises.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 conventional ACL reconstruction with quadruple flexor tendons and conventional physiotherapy (Active Comparator): This surgery is performed with the aid of videoarthroscopy in a minimally invasive manner. The procedure begins with the collection of the muscle graft that will be used for ACL reconstruction. The semitendinosus and gracilis muscles, also known as flexor tendons, will be used. All the participants will receive conventional physiotherapy with rehabilitation protocol with manual therapy, physical resources (heat, cold, electrotherapy), kinesiotherapy, and isokinetic exercises. All participants will be evaluated and re-evaluated in the same way.
  Interventions: Procedure: Group 1 ACL reconstruction with quadruple flexor tendons and conventional physiotherapy
- Group 2 (combined ACL + ALL reconstruction) and conventional physiotherapy (Active Comparator): Group 2 will undergo conventional ACL + ALL reconstruction in a similar manner to group 1 with quadruple flexor graft (triple semitendinosus and single gracilis). For combined ACL + ALL reconstruction, it is performed through a conventional tibial tunnel with a 55-degree angulation guide and a diameter defined by the thickness of the graft. All the participants will receive conventional physiotherapy with rehabilitation protocol with manual therapy, physical resources (heat, cold, electrotherapy), kinesiotherapy, and isokinetic exercises. All participants will be evaluated and re-evaluated in the same way.
  Interventions: Procedure: Group 2 ACL reconstruction with quadruple flexor tendons + ALL reconstruction

INTERVENTIONS:
Procedure: Group 1 ACL reconstruction with quadruple flexor tendons and conventional physiotherapy — Group 1 will undergo conventional ACL reconstruction with quadruple flexor tendons (double gracilis and semitendinosus). All the participants will receive conventional physiotherapy.
  Arms: Group 1 conventional ACL reconstruction with quadruple flexor tendons and conventional physiotherapy
Procedure: Group 2 ACL reconstruction with quadruple flexor tendons + ALL reconstruction — Group 2 will undergo conventional ACL reconstruction with quadruple flexor tendons (double gracilis and semitendinosus) + ALL reconstruction. All the participants will receive conventional physiotherapy.
  Arms: Group 2 (combined ACL + ALL reconstruction) and conventional physiotherapy

SUMMARY:
The objetive is compare knee joint stability, functional capacity, postural control, activation, and muscle strength of patients undergoing conventional Anterior Cruciate Ligament Reconstruction or the conventional Anterior Cruciate Ligament Reconstruction + Anterolateral Ligament Reconstruction technique of the knee, and rehabilitation for up to nine months. This project aims to include patients with ACL injuries already treated at the Knee Outpatient Clinic of the Hospital das Clínicas da UEL (HC-UEL), coordinated by the orthopedic physician Dr. Lucas da Fonseca Borghi, who has his master's degree related to this research project. Twenty patients between 18 and 50 years old, of both sexes, sedentary and/or active and/or athletes, diagnosed with unilateral injury of the Anterior Cruciate Ligament will be included. These patients will be evaluated, submitted to ACL surgery (conservative) or associated with ALL reconstruction and undergo rehabilitation with physiotherapy in conjunction with the extension project Sports Physiotherapy from Theory to Practice - Phase III (PROEX-UEL No 02675), coordinated by Prof. Dr. Christiane S. Guerino Macedo - advisor of this research. Expected results: It is expected that the group undergoing ACL + ALL reconstruction will present better knee joint stability, functional capacity, postural control, activation and muscle strength.

ELIGIBILITY:
Inclusion Criteria: - participants with 18 to 50 years old; - both sexes; - sedentary; -active; - athletes; - diagnosed unilateral ACL injury; - patients residing in the city of Londrina - PR.

Exclusion Criteria: - BMI (Body Mass Index) above 35 kg/m2; - multidirectional ligament laxity; - associated multiligament injury (PCL and posterolateral corner); - previous or current lower limb fractures; - previous ACL reconstruction (revision); - signs of osteoarthritis; - indication for meniscus suture; - neurological disease; - pregnant women; - heart disease; - previous lower limb surgeries.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Articular Range of Motion | preoperative and postoperative (5, 15, 30, 60 and 120 days).
  Assessment of hip and knee range of motion (Hip Internal Rotation Mobility and Lunge Test).
Functional Capacity | preoperative and postoperative (5, 15, 30, 60 and 120 days).
  Lysholm Knee Scoring Scale: Eight questions, with closed answer alternatives, whose final result is expressed in nominal and ordinal form.
Isometric Muscle Strength | preoperative and postoperative (5, 15, 30, 60 and 120 days).
  Dynamometer (SP MEDEOR/TECH), connecting it via Bluetooth to the My SP Tech application for verification to check the strength of knee flexors and extensors.

SECONDARY OUTCOMES:
Gait through the GaitRite program | postoperative 5, 15, 30, 60 and 10 days.
  Collection of spatiotemporal parameters related to the gait pattern in the pre and post-operative period using the GaitRite device. The GaitRite can help identify changes in knee loading, identify neuromuscular asymmetries, which may be caused by muscle weakness and identify movement patterns that may be causative of future injury or disability.
Functional Tests | preoperative and postoperative (5, 15, 30, 60 and 120 days).
  Star Excursion Balance Test: assess the dynamic stability of the lower limbs. The length of the participants' lower limbs will be measured to normalize the data obtained in each direction.
Analysis of postural control | preoperative and postoperative (5, 15, 30, 60 and 120 days).
  Will be tested on the BIOMEC411 force platform. The main balance parameters based on the center of pressure (COP) will be computed: the COP ellipse area (A-COP in cm2), average COP oscillation velocity (VEL in cm/s) in the anteroposterior (A/P) and mediolateral (M/L) movement directions, COP oscillation amplitude (cm) in the anteroposterior (A/P) and mediolateral (M/L) directions, and COP oscillation frequency (Hz) in the anteroposterior (A/P) and mediolateral (M/L) directions. All these variables are computed by the program based on the equilibrium parameters that the platform generates.
Analysis of muscle activation by surface electromyography | preoperative and postoperative (5, 15, 30, 60 and 120 days).
  The EMG signal will be captured with three pre-amplified active electrodes (gain: 1000) and filtered in a band-pass between 25 and 450 Hz, with a sampling frequency of 2000 Hz.

IPD SHARING:
Plan to Share IPD: Yes
Other researchers may contact us and request data from this research by email.
Supporting Information: CSR